CLINICAL TRIAL: NCT06692153
Title: A Multicenter, Pivotal, Randomized Controlled Trial Comparing the Safety and Efficacy of an Automated Insulin Delivery System With the Standard of Care in Adults With Type 2 Diabetes (EMBRACE-T2D)
Brief Title: Embecta AID System in Adults With Type 2 Diabetes
Acronym: EMBRACE-T2D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Program was discontinued.
Sponsor: Embecta Corp. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN202401
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Mellitus (T2DM); Type 2 DM; T2DM With Inadequate Glycemic Control; T2DM (Type 2 Diabetes Mellitus); T2D; T2DM
Keywords: AID system; AID; T2D; Type 2 Diabetes; Type 2 Diabetes Mellitus; IDD; Insulin Delivery Device; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Single Arm (Experimental): All participants will use the AID system.
  Interventions: Device: An AID System.
- Randomized Controlled Trial (RCT) (Experimental): Subjects will be randomized 2:1 in the AID group to SC group.
  Interventions: Device: An AID System.; Other: Standard of Care (SC)

INTERVENTIONS:
Device: An AID System. — The embecta Automated Insulin Delivery (AID) System is a closed loop system comprised of 3 components: the embecta insulin pump, a Smartphone with the Tidepool Loop app, and the Dexcom G6 CGM
Other: Standard of Care (SC) — Participants will continue to use their current therapy for T2D.
  Arms: Randomized Controlled Trial (RCT)

SUMMARY:
This is a multi-center, randomized control study that will evaluate the safety and effectiveness of the embecta Automated Insulin Delivery System in adults with Type 2 diabetes requiring insulin therapy

DETAILED DESCRIPTION:
This outpatient study consists of 2 phases.

Phase 1 (Single Arm) will establish the initial safety of the embecta AID system prior to initiating the phase 2 (RCT). Participants will follow the same protocol as the RCT AID group. During the treatment period all participants will undergo supervised exercise and meal challenges.

Phase 2 (Randomized Control Trial (RCT)) will be a 13-week parallel group RCT to evaluate the safety and efficacy with a 2:1 randomization to intervention with AID versus standard of care (SC) insulin therapy. The RCT AID group will use the embeca AID with Tidepool Loop app as well as the Dexcom G6 continuous glucose monitor (CGM).

Participants in both phases will do in-clinic or virtual visits at least monthly for a total of 9 visits. During the treatment period all participants will undergo supervised exercise and meal challenges.

ELIGIBILITY:
Key Inclusion Criteria:

1. Sufficient cognitive ability, per investigator judgment, to provide informed consent for study participation on an IRB approved consent form
2. ≥18 years of age at time of consent
3. Diagnosis of T2D, per investigator judgment, of at least 6 months duration prior to time of screening. Any permissible diabetes medications, including insulin, to the exclusion sulfonylurea, meglitinide, or repaglinides have been relatively stable for the past 30 days.
4. Currently treated with (1) multiple daily injections of insulin (MDI; defined as using basal insulin and at least one daily prandial injection), (2) an insulin pump without automation or (3) basal insulin without prandial insulin provided that screening HbA1c ≥7.5% (basal-only) for ≥3 months at the time of screening (per participant report and medical records available at the site)
5. Either not using any noninsulin glucose-lowering medications (such as GLP-1 receptor agonist, SGLT2 inhibitor, or other) or weight-reduction medications that can have a meaningful effect on glucose levels, or if using, then the dose has been stable for at least 4 weeks prior to screening based on investigator discretion
6. Willing to use U-100 (i.e., insulin lispro or insulin aspart) while using the embecta AID system if assigned to the AID group
7. Willing to not use concentrated insulin above U-100 or inhaled insulin while using the embecta AID system
8. Willing to participate in the study meal and exercise challenges if assigned to AID use in either the Single Arm Phase or the RCT AID group, and have a care partner, trained in hypoglycemia treatment guidelines including glucagon use, present during and immediately after the exercise challenges unless exercise challenges will be done in clinic.
9. Total daily insulin dose (TDD) <300 units/day
10. HbA1c ≤ 11% based on point-of-care or local lab measurement at screening
11. Willing to comply with study procedures, regardless of study arm
12. Able to read and understand English (due to user interface and IFU only being available in English)
13. Willing to have primary care provider and/or primary endocrinologist notified of participation in the trial
14. Investigator believes that the participant can successfully and safely operate all study devices and is capable of adhering to the protocol and completing the study
15. No medical, psychiatric, or other conditions, or medications being taken that in the investigator's judgement would be a safety concern for participation in the study. This includes considering the potential impact of medical conditions known to be present including cardiovascular, liver, kidney disease, thyroid disease, adrenal disease, malignancies, vision difficulties, active proliferative retinopathy, or other medical conditions; psychiatric conditions including eating disorders; drug or alcohol abuse
16. Participant is not capable of becoming pregnant, or if they are capable, they must meet one of the following criteria:

    a. has a negative urine pregnancy test and agrees to use one of the accepted contraceptive regimens throughout the entire duration of the trial from screening until last follow-up visit. The following contraceptive measures are considered adequate: i. Combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).

iii. Placement of an intrauterine device or intrauterine hormone- releasing system.

iv. Barrier methods of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository).

v. Has a vasectomized or sterile partner (where partner is sole partner of participant) and where vasectomy has been confirmed by medical assessment.

vi. Exercises true sexual abstinence. Sexual abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

or b. Participant is of non-childbearing potential due to menopause with at least one year since last menses or a medical condition confirmed by the investigator

Key Exclusion Criteria:

1. Use of an AID system within the last 3 months prior to screening
2. Use of systemic glucocorticoids within the last 8 weeks prior to screening or anticipated use of systemic glucocorticoids during the study (topical or inhaled or local injection into spine/joint -i.e., non-systemic is acceptable)
3. Current use of sulfonylurea, meglitinide, or repaglinides medications (within 30 days prior to screening)
4. Current use of hydroxyurea (within 1 day prior to screening) as hydroxyurea is known to cause falsely high CGM values which could lead to incorrect dosing from the AID system.
5. Has had more than 2 severe hypoglycemic events requiring third party help or hospitalization within the last 6 months prior to screening
6. Lack of reliable telephone service (for contact) or internet (smartphone containing the closed-loop algorithm application)
7. Planned surgery or hospitalization for which use of the embecta AID system would need to be discontinued for more than 7 days
8. Known allergy to medical grade adhesives that precludes use of the embecta AID system or CGM
9. Skin condition at the site(s) that may be used for application of the study CGM or embecta AID system that precludes use of the AID system or CGM
10. Dialysis planned or anticipated for chronic kidney disease in the next 4 months
11. Pregnant (positive urine hCG), breast feeding, plan to become pregnant in the next 2 months, or sexually active without use of contraception.
12. Current participation in another diabetes or obesity-related interventional clinical trial.
13. Anticipated change of residency or travel for more than 7 days at a time during the study that may, per investigator judgment, interfere with the completion of study visits, contacts, or procedures.
14. Immediate family member (spouse, biological or legal guardian, child, sibling, parent) of, or someone who is, an investigative site personnel directly affiliated with this study or who is an employee of embecta, Tidepool or the JAEB Center for Health Research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
HbA1c change | 13 weeks
  The change in HbA1c at 13 weeks from baseline

SECONDARY OUTCOMES:
CGM-measured time in range 70-180 mg/dL | 13 weeks
  Glucose metric from CGM
CGM-measured time in tight range 70-140 mg/dL | 13 weeks
  Glucose metric from CGM
CGM-measured time less than 54 mg/dL (non-inferiority, margin 0.5%) | 13 weeks
  Glucose metric from CGM
CGM-measured time less than 70 mg/dL (non-inferiority, margin 0.5%) | 13 weeks
  Glucose metric from CGM
CGM-measured mean glucose | 13 weeks
  Glucose metric from CGM
CGM-measured time greater than 180 mg/dL | 13 weeks
  CGM-measured time greater than 180 mg/dL
CGM-measured time greater than 250 mg/dL | 13 weeks
  Glucose metric from CGM
CGM-measured time less than 70 mg/dL | 13 weeks
  CGM-measured time less than 70 mg/dL
CGM-measured time less than 54 mg/dL | 13 weeks
  Glucose metric from CGM

OTHER OUTCOMES:
Safety - Severe hypoglycemia events | 13 weeks
  Severe hypoglycemia events as reported by PI
Safety - Diabetic ketoacidosis (DKA) events | 13 weeks
  Diabetic ketoacidosis (DKA) events as reported by PI
Safety - Hyperosmolar hyperglycemic (HHS) events | 13 weeks
  Hyperosmolar hyperglycemic (HHS) events as reported by PI
Safety - Other serious adverse events | 13 weeks
  Other serious adverse events as reported by PI
Safety - Unanticipated adverse device effects | 13 weeks
  Unanticipated adverse device effects as reported by PI
Safety - CGM-measured time less than 54 mg/dL | 13 weeks
  Glucose metric from CGM
Safety- CGM-measured hyperglycemia events | 13 weeks
  Glucose metric from CGM
Safety - CGM-measured hypoglycemia events | 13 weeks
  Glucose metric from CGM
Total daily insulin delivery | 13 weeks
  Insulin delivery metric from app
Percentage of insulin delivered as basal | 13 weeks
  Percentage of insulin delivered as basal
Weight change | 13 weeks
  Weight change from baseline to end of study as measured by PI
Type 2 Diabetes Distress Assessment System Core (T2-DDAS Core) | 13 weeks
  Type 2 Diabetes Distress Assessment System Core (T2-DDAS Core) as reported by participant
DAWN Impact of Diabetes Profile (DIDP) | 13 weeks
  DAWN Impact of Diabetes Profile (DIDP)
Diabetes Impact and Satisfaction (DIDS) Scale | 13 weeks
  Diabetes Impact and Satisfaction (DIDS) Scale as reported by participant
WHO-5 | 13 weeks
  WHO-5
Insulin Device Satisfaction Survey (IDSS) | 13 weeks
  Insulin Device Satisfaction Survey (IDSS) as reported by participant
Sleep Scale | 13 weeks
  Sleep Scale
System Usability Scale (SUS) | 13 weeks
  System Usability Scale (SUS) as reported by participant
Hypoglycemia Fear Survey II-Worry subscale only | 13 weeks
  Hypoglycemia Fear Survey II-Worry subscale only as reported by participant
EQ5D-5L | 13 weeks
  EQ5D-5L as reported by participant
Study-specific survey | 13 weeks
  Study-specific survey as reported by participant

CONTACTS AND LOCATIONS:
Overall Officials: Rayhan Lal, M.D., Study Chair — Stanford University
Locations (9):
- United States (9):
  - Stanford, Palo Alto, California
  - Diablo Research, Walnut Creek, California
  - Indiana Universtiy School of Medicine, Indianapolis, Indiana
  - NYC Research, Long Island City, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - UT Southwestern, Dallas, Texas
  - Tekton Research, Irving, Texas
  - Texas Diabetes & Endocrinology, Round Rock, Texas
  - DETS Utah, Sandy City, Utah